CLINICAL TRIAL: NCT07384871
Title: AI-Based Morphological Analysis and Biomechanical Numerical Evaluation of Mitral Valve Prolapse (MVP) From Real-Time 3D Echocardiography (RT3DE)
Brief Title: AI-Based Shape and Function Analysis of Mitral Valve Prolapse Using 3D Ultrasound
Acronym: AI4MVP
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Sponsor
Other Study IDs: AI4MVP
Record Dates: First submitted 2026-01-12; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Mitral Valve Prolapse; Myxomatous Mitral Valve Degeneration
MeSH Terms: conditions — Mitral Valve Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — In case of surgically excised MV tissue due to substantial (i.e., at least 10×10 mm) leaflet resection, samples of leaflets' tissue will be harvested and therefore stored in the institutional BioCor biobank for subsequent histomorphometric analysis. Collected samples will undergo quantitative analysis of tissue thickness and ad hoc structural stains of leaflet morphological features. Biological samples will be finally destroyed after the evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop and validate a fully automated imaging and modeling pipeline for the analysis of mitral valve prolapse (MVP) using real-time three-dimensional transesophageal echocardiography (RT3DE). The primary goal is to automatically segment mitral valve (MV) substructures, extract anatomical landmarks, and generate 3D models of the MV apparatus to characterize morphological and functional features of degenerative MVP. Advanced deep learning techniques and geometric processing tools will be applied to enable automated analysis.

A secondary objective is to build patient-specific finite element (FE) models based on RT3DE data to evaluate the biomechanical consequences of MVP and to simulate the effects of surgical repair. These simulations will assess stress distribution and force transmission within the MV apparatus.

Additionally, in cases where substantial surgical resection of MV tissue occurs, excised leaflet samples will be collected and preserved for histological and morphometric analysis.

DETAILED DESCRIPTION:
This prospective study aims to investigate the anatomical and biomechanical characteristics of MVP using RT3DEE and advanced artificial intelligence (AI)-based image analysis techniques. The goal is to develop an automated framework for the segmentation and morphological assessment of the MV apparatus, and to conduct FE modeling to evaluate the biomechanical implications of degenerative MVP and associated surgical repairs.

Imaging Protocol Intraoperative RT3DE will be performed in the operating room as part of the standard imaging protocol during surgical MVP repair. A Vivid S70N ultrasound system (GE Healthcare) equipped with a 6VT 4D multiplane RT3DE probe will be used. Standard mid-esophageal RT3DE views will be acquired, including full left ventricular (LV) chamber volumes and zoomed, gated 3D views of the MV complex (annulus, leaflets, and papillary muscles). To enhance image quality, zoomed acquisitions will be limited to the smallest pyramidal volume capturing the entire mitral complex, ensuring frame rates ≥20 Hz. All imaging datasets will be anonymized prior to analysis.

Surgical Protocol MVP surgical repair will be conducted under general anesthesia through a right mini-thoracotomy. Surgical techniques will include: i) leaflet resection (removal of excess leaflet tissue); ii) neochordal implantation (placement of expanded polytetrafluoroethylene, ePTFE, artificial chordae); annuloplasty (implantation of an annuloplasty ring or pericardial band for annular stabilization).

In cases where significant leaflet tissue is excised (≥10×10 mm), samples will be collected and stored in the institutional BioCor biobank for histological and morphometric analysis. Samples will be decontaminated, cryopreserved, and stored at -80°C. After histological evaluation, all biological material will be destroyed.

Clinical Data Collection Demographic (e.g., age, sex) and clinical data (e.g., diagnosis, medications, comorbidities) will be obtained from medical records and anonymized.

Neural Network Training for Image Segmentation Anonymized RT3DE datasets will be manually segmented by expert operators using advanced image analysis software (e.g., 3D Slicer). A minimum of 150 RT3DE acquisitions will be processed to generate binary masks of the MV annulus, leaflets, and papillary muscles.

These segmented datasets will be used to train a convolutional neural network (CNN), likely based on the 3D U-Net architecture; 70% of the datasets will be used as training data and 30% will be reserved for testing and validation.

The CNN will learn to automatically segment MV structures and generate 3D surface models. Key anatomical features-such as annulus contour, leaflet free margin, commissures, and papillary muscle positions-will be extracted automatically.

Quantitative geometric parameters will include annular area, perimeter, anteroposterior diameter, commissural width, annular height and ellipticity, leaflet dimensions, coaptation zones and billowing extent.

FE Analysis Patient-specific 3D models of the mitral valve will be reconstructed from the segmented RT3DE data. These models will undergo smoothing and remeshing to generate high-quality meshes for structural FE analysis. Chordae tendineae will be modeled based on established anatomical templates and tuned to match physiological lengths. Tissue material properties will be assigned based on published experimental data.

FE simulations will be used to quantify stress distribution on MV leaflets, assess load transfer between leaflets and papillary muscles and evaluate mechanical effects of surgical interventions (e.g., neochordal implantation, annuloplasty) These simulations are retrospective and exploratory; they will not influence surgical decision-making.

Follow-up No post-operative follow-up is required beyond standard clinical care. The study is focused on intraoperative imaging and tissue collection, followed by offline image analysis and computational modeling.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 years old);
* Documented symptomatic degenerative MR with indication to MVP surgical repair, following the Heart Team decision;
* Periprocedural transesophageal 3DRTE of the MV apparatus, which is clinical standard modality for morphological assessment and guidance during MVP surgical repair;
* Signed informed consent.

Exclusion Criteria:

* Inadequate quality of 3DRTE imaging, e.g., due to inadequate patient-specific acoustic window;
* 3DRTE imaging with a temporal resolution of < 20 Hz;
* Patient treated through prosthetic MV replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will focus on patients referred to IRCCS Policlinico San Donato for surgical MVP repair. The study will exploit the standard clinical imaging required during MVP surgical repair and will have no impact on the clinical procedure. No variation in prophylaxis or follow-up is expected compared to those of practice as suggested by the international guideline. Hence, there are no physical, psychological, and social risks and/or direct benefits associated with the activities carried out during the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Accuracy of automated MV substructure segmentation and extraction of anatomical landmarks from RT3DE | 36 months
  The accuracy of AI-based automated segmentation of MV substructures (anterior and posterior leaflets, mitral annulus, and papillary muscles) from RT3DE is assessed using expert manual segmentation as reference standard and analyzing the following measures: i) Dice Similarity Coefficient (DSC, -); ii) Mean Surface Distance (MSD, mm); iii) Hausdorff Distance (HD, mm). Accuracy of AI-based automated identification of key MV anatomical landmarks relevant to degenerative mitral valve prolapse is assessed compared with expert manual annotation analyzing the Euclidean distance error (mm) between automated and expert-defined landmarks (annular hinge points, leaflet free-edge points, coaptation line, papillary muscle tips).

SECONDARY OUTCOMES:
Automated quantification of MV morphometric and functional descriptors | 36 months
  Ability of the automated pipeline to derive consistent quantification - compared to commercially available solutions for RT3DE processing - of clinically relevant morphometric and functional descriptors of degenerative MVP from RT3DE: i) mitral annular dimensions (projected area, mm²; perimeter, mm; antero-posterior and commissural diameters, mm; height, mm; ellipticity, -); ii) leaflet surface area and billowing volume (mm², mm³); leaflet prolapse height and prolapse volume (mm, mm³); coaptation length and coaptation area (mm, mm²).
Change in mechanical stress of MV leaflets following surgical MVP repair | Up to 1 month after MVP surgical repair
  Assessment of change in mechanical stress of MV leaflets following surgical MVP repair using patient-specific FE MV models derived from RT3DE, comparing peak and mean leaflet stress (kPa) between degenerative MVP and post-repair conditions.
Change in mechanical load transfer to MV sub-apparatus following surgical MVP repair | Up to 1 month after MVP surgical repair
  Assessment of changes in the mechanical load transfer to MV sub-apparatus following MV surgical repair using patient-specific FE MV models derived from RT3DE, comparing chordal forces and load transfer to MV papillary muscles (N) between degenerative MVP and post-repair conditions.
Change in mechanical stress of MV papillary muscles following surgical MVP repair | Up to 1 month after MVP surgical repair
  Assessment of change in mechanical stress acting on MV papillary muscles following surgical MVP repair using patient-specific FE MV models derived from RT3DE, comparing peak and mean stress (kPa) between degenerative MVP and post-repair conditions.
Change in coaptation of MV leaflets following surgical MV repair | Up to 1 month after MVP surgical repair
  Assessment of change in MV leaflet coaptation following surgical MVP repair using patient-specific FE MV models derived from RT3DE, comparing coaptation length and area (mm, mm²) between degenerative MVP and post-repair conditions.
Thickness of MV leaflet tissue excised during MVP surgical repair | Up to 2 weeks after MVP surgical repair
  Assessment of the thickness (mm) of MV leaflet tissue excised as a consequence of substantial leaflet resection during surgical MVP repair.
Degree of myxomatous degeneration of excised MV leaflet tissue | Up to 2 weeks after MVP surgical repair
  Gross and histomorphometric assessment of the degree of myxomatous degeneration of MV leaflet tissue surgically excised during MVP surgical repair, using a semi-quantitative score (0-3): 0 = absent (no gross or histological evidence); 1 = mild (limited focal myxoid/proteoglycan extracellular matrix expansion with mild collagen disorganization); 2 = moderate (diffuse or multifocal myxoid/proteoglycan expansion with moderate collagen fragmentation/disorganization and leaflet thickening); 3 = severe (extensive/diffuse myxoid degeneration with marked extracellular matrix expansion, severe collagen disruption, and pronounced leaflet thickening/redundancy).
Structural histological analysis of excised myxomatous MV leaflet tissue | Up to 2 weeks after MVP surgical repair
  Quantitative histological assessment of myxomatous degeneration of excised MV leaflet tissue obtained during mitral valve prolapse (MVP) surgical repair, quantifying collagen and elastin content (% of tissue area) through structural stains.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Italy